CLINICAL TRIAL: NCT04399746
Title: A Pilot Study for COVID-19 Outpatient Treatment With the Combination of Ivermectin-azithromycin-cholecalciferol
Brief Title: Ivermectin-Azithromycin-Cholecalciferol (IvAzCol) Combination Therapy for COVID-19
Acronym: IvAzCol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Guadalupe Espitia Hernandez, MD, PhD, Investigator, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IvAzCol
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: COVID
MeSH Terms: interventions — Ivermectin; Azithromycin; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Relation 3:1 in Combination:Control groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination (Experimental): Ivermectin (6mg once daily in day 0,1,7 and 8) plus Azithromycin (500mg once daily for 4 days) plus Cholecalciferol (400 IU twice daily for 30 days).
  Interventions: Drug: Ivermectin; Drug: Azithromycin; Drug: Cholecalciferol
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Ivermectin — 6mg once daily in day 0,1,7 and 8
  Arms: Combination
Drug: Azithromycin — 500mg once daily for 4 days
  Arms: Combination
Drug: Cholecalciferol — 400 IU twice daily for 30 days
  Arms: Combination

SUMMARY:
As the world faces COVID-19, the search for effective treatments against the disease and its complications has turned its gaze to drugs that are classically used in other infectious diseases. Some drugs are being examined for the recent evidence on its effects on viral replication and inflammation, one is Azithromycin, used to treat a wide variety of bacterial infections, Ivermectin, an anti-parasitic drug and the other is Cholecalciferol to increase serum concentration of 25-hydroxyvitamin D.

DETAILED DESCRIPTION:
The aim of the study is to assess the efficacy of Ivermectin-Azithromycin-Cholecalciferol combination in COVID-19 in early stages of the disease with outpatient management.

Enrollment of subject into the trial shall only occur after providing written permission to voluntarily participate into the study by signing and dating the informed consent form before starting any trial related treatment. 30 cases of COVID-19 will be enrolled into the trial with a 3:1 proportion, divided into two groups. First group with confirmed cases of COVID-19 shall be treated with Ivermectin (6mg once daily in day 0,1,7 and 8) plus Azithromycin (500mg once daily for 4 days) plus Cholecalciferol (400 IU twice daily for 30 days) in an outpatient regimen. The second group with confirmed cases of COVID-19 who refused treatment were shall be allocated as the control group for monitoring.

Test for virus at day 1 and 14 from beginning of trial drug started for the outpatient regimen.

Clinical symptoms, oxygen saturation and oxygenation index will be monitored every day of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed infection of SARS-CoV2 virus
* Mild COVID-19
* Symptoms of respiratory illness
* Cough
* Fever (T >38 °C)

Exclusion Criteria:

* Allergy to any of the drugs treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Viral clearance | 14 days
  Test for virus at day 1 and 14 from beginning of trial drug started

SECONDARY OUTCOMES:
Symptoms duration | 14 days
  The duration of symptoms in days
SpO2 | 14 days
  oxygen saturation
SpO2/FiO2 | 14 days
  Oxygen Saturation (SpO2)/Fraction of Inspired Oxygen (FiO2) Ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient treatment, Mexico City, Mexico